CLINICAL TRIAL: NCT01357603
Title: A Randomized, Double-blind, Two Period, Cross Over Glucose Clamp Study to Test for Bioeqivalence Between Two Long Acting Insulin Analogs-Wockhardt's Glaritus™ (Insulin Glargine) and Lantus (Insulin Glargine) in Subjects With Type 1 Diabetes
Brief Title: Comparative Glucose Clamp Study of Wockhardt's Recombinant Insulin Analog Glargine(Glaritus) With Lantus in T1DM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wockhardt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: Glaritus/PK-PD/FDA/2011
Record Dates: First submitted 2011-05-12; First posted 2011-05-20 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Type1 Diabetes
MeSH Terms: interventions — Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glaritus arm (Experimental): Insulin glargine (Glaritus: 100 U/ml), Penfill® cartridges 3.0ml
  Interventions: Biological: Glargine
- Lantus arm (Active Comparator): Insulin glargine (Lantus: 100 U/ml), Penfill® cartridges 3.0ml
  Interventions: Biological: Glargine

INTERVENTIONS:
Biological: Glargine — dosage form: Subcutaneous injection

SUMMARY:
The aim of this trial is to demonstrate bioequivalence of Glaritus® to Lantus® with regard to its total and to its maximum serum insulin concentrations.

DETAILED DESCRIPTION:
The purpose of this study is to test for bioequivalence based on the pharmacokinetic parameter AUC INS-GLR 0-24h and on pharmacodynamic parameter AUC GIR 0-24h between the two long-acting insulin glargine formulations, Lantus® and Wockhardt's Glaritus® in subjects with type1 diabetes as well as assessing safety and local tolerability of the two insulin preparations.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects with type 1 diabetes ≥12 months.
2. HbA1c ≤9% by local laboratory analysis (one retest within a week is permitted with the result of the last test being conclusive).
3. Age ≥18 and ≤60 years.
4. Considered generally healthy upon completion of medical history, physical examination and biochemical investigations as judged by the Investigator.
5. Signed and dated informed consent obtained before any trial-related activities. (Trial-related activities are any procedure that would not have been performed during normal management of the subject).

Exclusion Criteria:

1. Previous participation in this trial, or participation in other clinical trials within the last 30 days.
2. Pregnant, breast-feeding or the intention of becoming pregnant or not using adequate contraceptive measures (e.g. intrauterine device (IUD) that has been in place for at least 3 months, or sterilization, or the oral contraceptive pill, which should have been taken without difficulty for at least 3 months, an approved hormonal implant or double barrier method including male condoms used plus spermicide, diaphragm with spermicide plus male condom, cap with spermicide plus male condom).
3. History of any illness that, in the opinion of the Investigator, might confound the results of the trial or pose risk in administering the trial drug to the subject. In particular, subjects with significant cardiovascular disease, anemia (hemoglobin below the lower limit of normal) or hemoglobinopathy will not be allowed to enter the trial.
4. Cardiac problems defined as decompensated heart failure (New York Heart Association (NYHA) class III and IV) at any time and/or angina pectoris within the last 12 months and/or acute myocardial infarction at any time.
5. Clinically significant abnormal ECG at screening, as judged by the Investigator.
6. History of alcohol or drug abuse in the past five years.
7. Any positive reaction of drug abuse.
8. Hepatitis B or C or HIV positive.
9. Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.
10. History of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reaction.
11. Regular cigarette smoker, defined as smoking >1 pack/day and unable to refrain from smoking during the in house period.
12. Known or suspected allergy to trial product or related products.
13. Any disease or condition that, in the opinion of the Investigator, would represent an unacceptable risk for the subject's safety.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 111 (Actual)
Dates: Start 2011-06; Primary Completion 2012-05 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Pharmacokinetic parameter:AUC INS-GLR 0-24h. | over 24hrs post dose
Bioequivalence based on Pharmacodynamic parameter: AUC GIR 0-24hrs | over 24hrs post dose
Pharmacokinetic Parameters: Maximum concentration (Cmax) | over 24hrs post dose

SECONDARY OUTCOMES:
Safety parameters | till 24 hrs post-dose
  Number of AE's, SAE's, Hypoglycemic events and local tolerability
Pharmacodynamic parameters: Area under curve glucose infusion rate from 0-24hrs | over 24hrs post dose
  AUC GIR 0-12h,AUC GIR 12-24h,AUC GIR 0-24h
Pharmacokinetic parameter: Area under curve from 0-24hrs | over 24hrs post dose
  AUC INS-GLR 0-12hrs, AUC INS-GLR 12-24hrs,AUC INS-GLR 0-24hrs
Pharmacokinetic Parameters: tmax and t1/2 | over 24hrs post dose
Pharmacodynamic parameter: GIR max and tGIR max | over 24hrs post dose

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Elaine Watkins, Principal Investigator — Profil Institute of Clinical Research
Locations (1):
- Profil Institute for clinical Research, Chula Vista, California, United States